CLINICAL TRIAL: NCT02553629
Title: Effect of Depth of Neuromuscular Block on Intraoperative Surgical Conditions as Determined by the Leiden Surgical Rating Scale in Morbidly Obese Patients Undergoing Laparoscopic Bariatric Surgery
Brief Title: Effect of Deep Neuromuscular Block on Surgical Conditions in Morbidly Obese Patients
Acronym: BLISS3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Medical Center Haaglanden (Other)
Responsible Party: Principal Investigator, Albert Dahan, MD, PhD, professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL52829.058.15
Record Dates: First submitted 2015-08-28; First posted 2015-09-17 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Surgical Conditions
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- moderate neuromuscular block (Active Comparator): rocuronium 0.1-0.6 mg/kg aimed at a train of four of 1 - 2 twitches
  Interventions: Drug: Rocuronium
- deep neuromuscular block (Experimental): rocuronium 0.1-0.6 mg/kg aimed at a post tetanic count of 1 - 2 twitches
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium

SUMMARY:
This is a randomized control trial (RCT) that studies the surgical conditions during moderate and deep neuromuscular blockade in 100 morbidly obese patients receiving elective laparoscopic surgery for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* BMI > 34 kg/m2
* Elective bariatric surgery.

Exclusion Criteria:

* Known or suspected neuromuscular disorders impairing neuromuscular function
* Allergies to muscle relaxants, anesthetics or narcotics
* A(family) history of malignant hyperthermia
* Women who are or may be pregnant or are currently breast feeding
* Renal insufficiency, as defined by serum creatinine x 2 of normal, or urine output < 0.5 ml/kg/h for at least 6 h.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD, PhD, professor, Principal Investigator — LUMC
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - Medisch Centrum Haaglanden / Nederlandse Obesitas Kliniek, The Hague, South Holland

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Neuromuscular Block: rocuronium 0.1-0.6 mg/kg aimed at a train of four of 1 - 2 twitches
  Rocuronium
- Deep Neuromuscular Block: rocuronium 0.1-0.6 mg/kg aimed at a post tetanic count of 1 - 2 twitches
  Rocuronium
Period: Overall Study
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Started | 53 | 56
Completed | 50 | 50
Not Completed | 3 | 6
Not completed — Logistic reasons | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (10.6) | 47.2 (11.1) | 47.1 (10.9)
Gender [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Surgical Rating
Description: During a procedure, the surgical condition will be scored by one surgeon using a 5-point surgical rating. This will be done at 10 min intervals from the start of surgery until the end of surgery scale. The rating scale is a 5-point ordinal scale ranging from 1 = poor condition to 5 = optimal surgical conditions. The mean difference in ratings between procedures under deep neuromuscular block and those during moderate neuromuscular block will be evaluated.
  The rating scale will be averaged for each subject and the mean values will be reported.
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 50 | 50
units on a scale | 4.2 (0.7) | 4.8 (0.2)
Statistical Analysis 1: Comparison: Moderate Neuromuscular Block vs Deep Neuromuscular Block; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis

2. Secondary Outcome: Extubation
Description: The investigators will assess the time from the injection of the reversal agent until the time to removal of the endotracheal tune (extubation).
Time Frame: intraoperative
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 50 | 50
minutes | 3 [1 to 6] | 3 [1 to 8]
Statistical Analysis 1: Comparison: Moderate Neuromuscular Block vs Deep Neuromuscular Block; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

3. Secondary Outcome: Pain
Description: pain will be scored using numeric rating scale (0-10, with 0 = no pain and 10 = most pain imaginable), at 10 minute intervals at the post anesthesia care unit, but only the mean value will be used in the analysis and reported.
Time Frame: postoperative, for up to 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 50 | 50
units on a scale | 4.4 (1.4) | 3.9 (1.4)
Statistical Analysis 1: Comparison: Moderate Neuromuscular Block vs Deep Neuromuscular Block; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

4. Secondary Outcome: Respiration
Description: Respiration will be measured by counting the respiratory rate at 10 min interval for 2 hours in the post anesthesia care unit. The breaths per min (unit 1/min) will be logged.
  The data were averaged per subject and the mean of the mean data are reported.
Time Frame: 2 hours postoperative
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 50 | 50
breaths per minute | 12.7 (0.7) | 12.6 (1.1)
Statistical Analysis 1: Comparison: Moderate Neuromuscular Block vs Deep Neuromuscular Block; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

5. Secondary Outcome: Mean Arterial Blood Pressure
Description: Mean arterial pressure (MAP in mmHg) will be monitored at 10 minute intervals for 2 hours in the post anesthesia care unit.
  The data will be averaged per subject and the mean of the mean values are reported.
Time Frame: 2 hours postoperative
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Number analyzed (Participants) | 50 | 50
millimeters of mercury | 98 (13) | 101 (15)
Statistical Analysis 1: Comparison: Moderate Neuromuscular Block vs Deep Neuromuscular Block; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Moderate Neuromuscular Block | Deep Neuromuscular Block
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No